CLINICAL TRIAL: NCT03807297
Title: Comparative Study Between TIVA Vs Inhalational Modes of Anaesthesia in Patients Undergoing Modified Radical Mastectomy
Brief Title: TIVA vs Inhalational Mode of Anaesthesia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rajiv Gandhi Cancer Institute & Research Center, India (Other)
Responsible Party: Principal Investigator, Dr. Nitesh Goel, Dr. Nitesh Goel - Consultant Anaesthesia, Rajiv Gandhi Cancer Institute & Research Center, India
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: RajivGCIRC2
Record Dates: First submitted 2019-01-05; First posted 2019-01-16 (Actual); Last update posted 2020-02-19 (Actual); Status verified 2020-02

CONDITIONS: Anesthesia Awareness
Keywords: total intravenous anesthesia
MeSH Terms: conditions — Intraoperative Awareness | interventions — Injections; Propofol; Sevoflurane; Nitrous Oxide

STUDY DESIGN:
Intervention Model Description: two groups - one for Total Intravenous Anaesthesia mode and other for Inhalational mode of anaesthesia
Who Masked: Participant, Investigator
Masking Description: participants will be alloted in two groups as per chit system and won't be aware of type of anaesthesia, investigator won't be aware of type of anaesthesia and will record the data.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- TIVA - total intravenous anaesthesia (Other): only intravenous type of anaesthesia using Injection propofol, 10 mg and Injection dexmedetomidine drug infusion will be infused for maintenance of anaesthesia
  Interventions: Drug: Injection dexmedetomidine; Drug: Injection, Propofol, 10 Mg
- Inhalational anaesthesia (Other): In this group, both nitrous oxide and sevoflurane will be given for maintenance of anaesthesia
  Interventions: Other: sevoflurane; Other: nitrous oxide

INTERVENTIONS:
Drug: Injection dexmedetomidine — alpha 2 a agonist used for sedation, analgesia
  Other Names: dexmed
  Arms: TIVA - total intravenous anaesthesia
Drug: Injection, Propofol, 10 Mg — non barbiturate type of intravenous anaesthetic drug
  Other Names: propofol spiva
  Arms: TIVA - total intravenous anaesthesia
Other: sevoflurane — inhalational anaesthetic agent
  Arms: Inhalational anaesthesia
Other: nitrous oxide — inhalational anaesthetic agent
  Arms: Inhalational anaesthesia

SUMMARY:
Sevoflurane based inhalational anaesthesia is the preferred mode of anesthesia for small duration cases. But in recent times, concept of rapid discharge, day care procedures, and green environment has created the need of new modalities of anaesthesia for such cases. Considering such factor, investigators have planned using TIVA i.e. total intravenous anaesthesia with Inj. Propofol and Inj. Dexmedetomidine infusions for maintenance of anesthesia in Modified Radical Mastectomy (MRM). By comparing the two modalities of anaesthesia i.e. TIVA vs Inhalational investigators are trying to find out whether TIVA is feasible, cost effective and comparable to inhalational anaesthesia in terms of intraoperative hemodynamic stability, pain, intraoperative awareness and recovery profile. This comparison and analysis will help to determine if TIVA can be used as the sole mode of anaesthesia during MRM as it will initiate early discharge of patient and will contribute to the Green OT concept.

DETAILED DESCRIPTION:
Aim: To compare TIVA Vs Inhalational mode of anaesthesia in patients undergoing Modified Radical Mastectomy

Objective:

* Feasibility of TIVA in Modified Radical Mastectomy
* Cost - effectiveness of TIVA Vs Inhalational anesthesia
* Effectiveness of TIVA as compared to Inhalational Anaesthesia by comparing intraoperative hemodynamic parameters and recovery profile.

Study design: It will be a prospective randomized controlled interventional type of study.

Sample size: Total 100 patients will be recruited for two groups i.e. 50 each in -TIVA (T) and Inhalational (I) group. Groups will be allocated as per chit system to remove the bias.

In group T: (TIVA): Inj. Dexmedetomidine will be started at induction @1mcg/kg over 10 min followed by 0.2 to 0.7 mcg/kg/hr along with propofol @ 75mcg/kg/min (25-100 mcg/kg/min) for maintenance of anaesthesia.

In group I: (inhalational): both nitrous oxide (in ratio of 50:50 with oxygen) and sevoflurane will be started at induction.

In both groups drugs and gases (respective to groups) will be titrated to maintain a bispectral index value between 40-60. Anaesthetic drugs will be stopped at last skin suture. Soon after reversal- recovery profile, modified Aldrete score will be recorded along with time taken to first eye opening and attainment of BIS value of >90. At the end of case amount of each agents consumed will be recorded - i.e. nitrous oxide, sevoflurane, propofol, dexmedetomodine- for cost analysis.

ELIGIBILITY:
Inclusion Criteria:

* Age group: 30-65 yrs
* ASA status: 1-3
* Use of endotracheal tube for securing the airway

Exclusion Criteria:

* CKD, CLD patients
* Cardiac dysfunction
* Psychotic and neurotic disorders
* Drug addiction
* BMI > 30
* Use of supraglottic device
* Use of any nerve blocks

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2019-01-10 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
total intravenous anesthesia | 3 hours
  Intraoperative Bispectral index maintenance between 40-60

SECONDARY OUTCOMES:
Cost - effectiveness | 3 hours
  cost of drugs consumed per patient in both groups

CONTACTS AND LOCATIONS:
Overall Officials: NITESH GOEL, MBBS,DA,DNB, Principal Investigator — Rajiv Gandhi Cancer Institute And Research Centre
Locations (1):
- Rajiv Gandhi Cancer Institute and Research Centre, New Delhi, National Capital Territory of Delhi, India